CLINICAL TRIAL: NCT00808223
Title: A Phase 2, Single-Arm Study to Evaluate the Safety and Pharmacokinetics of Alefacept in Adolescent Subjects With Moderate to Severe Psoriasis [ISN 0485-CL-0004]
Brief Title: Safety and Pharmacokinetics (PK) of Alefacept in Adolescent Subjects With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0485-CL-0004; 2008-005830-63 (EudraCT Number)
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Psoriasis
Keywords: alefacept; adolescent; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1. alefacept (Experimental)
  Interventions: Biological: alefacept

INTERVENTIONS:
Biological: alefacept — IM injection
  Other Names: Amevive; ASP0485

SUMMARY:
To establish the safety of alefacept when administered to adolescent subjects with moderate to severe psoriasis.

DETAILED DESCRIPTION:
A planned interim analysis will be conducted to evaluate safety and pharmacokinetics following the Week 4 evaluation of approximately the first 12 subjects. A dose adjustment may be implemented based on these results. A preliminary review of the Week 4 pharmacokinetics of the first 6 subjects will occur to monitor exposure. If a dose adjustment is required, pharmacokinetics will be repeated for the first 12 subjects enrolled at the new dose (subjects 13-24).

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate to severe chronic plaque psoriasis involving at least 10% or greater body surface area
* Subject is a candidate for systemic treatment or phototherapy
* Subject is in good health and alefacept is not contraindicated
* Subject must have absolute total CD4+ lymphocyte counts within the normal range at screening
* Female subjects of child bearing potential have a negative pregnancy test prior to first dose of alefacept and agree to practice effective contraception during the study
* Subject must have predosing laboratory findings without clinically significant abnormal values for hematocrit, hemoglobin, platelets, white blood count and differential, serum creatinine, bilirubin, ALT, AST and prothrombin.
* Subject must have completed all standard childhood immunizations at least 12 weeks prior to the first dose
* Subject meets medication washout requirements and agrees to follow medication restrictions during the study
* Subject agrees to comply with the study requirements and agrees to come to the clinic for required study visits

Exclusion Criteria:

* Subject has a primary dermatological diagnosis of psoriasis other than plaque psoriasis
* Subject has a known hypersensitivity to alefacept or any excipient of the study medication
* Subject has had a serious local infection or systemic infection within 12 weeks prior to the first dose of study drug
* Subject has a fever (body temperature ≥ 38°C [or > 37°C for sites in Latvia]) or symptomatic viral or bacterial infection (including upper respiratory tract infection) within 1 week prior to the first dose of study drug
* Subject is known to be positive for HIV antibodies
* Subject has a history of chronic serious infection including hepatic disease or has positive result to serology test for hepatitis A antibody IgM, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) antibody or, in Europe, tubercle bacillus (TB) at Screening
* Subject has a history or evidence of tuberculosis based on serology or a positive PPD skin test at Screening
* Subject has had treatment with any immunosuppressant agent within 12 weeks, any antibody or immuno-globulin within 24 weeks, or any investigational drug or approved therapy for investigational use within 8 weeks prior to the first dose of study drug
* Subject has had more than six herpes simplex virus (HSV) breakouts per year or is currently having an outbreak or has had an outbreak within the last 24 weeks
* Subject has a history of malignancy (other than non-melanoma skin cancers)
* Subject has a chronic condition which is not well controlled
* Subject is pregnant or nursing
* Subject has a history of severe allergic or anaphylactic reactions

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assessment of Physical exams, vital signs, select blood chemistry and hematology, lymphocyte subset analysis, anti-alefacept antibody monitoring, adverse event monitoring including infections. | 6 months

SECONDARY OUTCOMES:
Assessment of Pharmacodynamics: Total lymphocytes and lymphocyte subsets | 4 Weeks
Assessment of Pharmacokinetics through analysis of blood samples (only approximately first 24 subjects enrolled) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Medical Affairs, Study Director — Astellas Pharma Global Development
Locations (5):
- United States (2):
  - Pediatric and Adolescent Dermatology, San Diego, California
  - Physicians Skin Care, PLLC, Louisville, Kentucky
- First Municipal Hospital for Active Treatment - Sofia, Sofia, Bulgaria
- Latvia (2):
  - Skin and STD Clinical Centre, Riga
  - Department of Dermatology No.17, Children Clinical Hospital, Riga